CLINICAL TRIAL: NCT03577496
Title: Does Aromatherapy Decrease Postoperative Nausea and Vomiting?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-0058
Record Dates: First submitted 2018-06-23; First posted 2018-07-05 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-06

CONDITIONS: Nausea, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — peppermint oil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peppermint oil (Experimental): A cotton ball with three drops of peppermint oil will be waved under the patient's nares upon arrival to the recovery room. The patients will be assessed for PONV for up to an hour in the post anesthesia care unit (PACU) or until their discharge, whichever is first.
  Interventions: Other: Peppermint oil

INTERVENTIONS:
Other: Peppermint oil — A cotton ball with three drops of peppermint oil will be waved under the patient's nares.

SUMMARY:
Aromatherapy has been proven to be effective for treating patients with postoperative nausea and vomiting (PONV) after surgery, but few studies analyze its effect on preventing PONV. Most studies use aromatherapy once patients become nauseous, but this study will address a gap in the literature with relation to the effect of aromatherapy in the prevention of PONV.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine if aromatherapy will prevent postoperative nausea and vomiting (PONV). Peppermint aromatherapy will be used preemptively to test for effectiveness, decreased PONV, and the ability to avoid anti-emetics. This study will seek to demonstrate that peppermint aromatherapy is a simple, cost effective way to prevent PONV after anesthesia. By decreasing the need for anti-emetics and incidence of PONV, patients may have a quicker recovery time and experience less side effects from anti-emetics, such as increased sedation. This problem is significant to patients and society as it may demonstrate that the inhalation of peppermint can ease PONV and decrease costs due to anti-emetics, wound dehiscence, and prolonged hospital stay. This study may lead to higher levels of patient satisfaction; if the patients are not nauseated they may be more satisfied with their care.

ELIGIBILITY:
Inclusion Criteria:

* Adult surgical patients ages 18 and older.
* Patients deemed medically stable by their surgery team.
* Anesthesia and Surgeon faculty approval will be obtained prior to asking the patient for their consent.

Exclusion Criteria:

* Minors
* Unstable patients, such as ICU patients or intubated patients, pregnant women, and prisoners.
* Patients with a history of severe PONV or severe delirium on emergence from anesthesia will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Decrease incidence of postoperative nausea and vomiting (PONV) | Patients will be monitored for up to one hour after surgery to test effectiveness of peppermint oil at decreasing PONV.
  Decreased severity of PONV rating with peppermint aromatherapy

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Karsten, RN, BSN, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided